CLINICAL TRIAL: NCT04368468
Title: Study of the Modifications of the Immune Microenvironment Induced by Neoadjuvant Chemotherapy in Triple-negative Breast Cancers
Brief Title: Modifications of Immune Microenvironment Induced by Neoadjuvant Chemotherapy in Triple-negative BC
Acronym: MIMOSA
Status: Completed | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Other Study IDs: 19HLSEIN02
Record Dates: First submitted 2020-04-20; First posted 2020-04-29 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Triple Negative Breast Cancer
Keywords: post neo adjuvant therapy; immune micro environment; biomerker chacterization
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — microbiopsy of the breast primary tumor preserved in FFPE and of the operative part preserved in FFPE.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: biomarker evolution — analysis of a list of biomarkers on triple negative breast tumors samples before and after neoadjuvant therapy
  Other Names: triple negative breast cancer biomarker evolution

SUMMARY:
The prescription of neoadjuvant chemotherapy becomes a standard in women with HER2-positive or triple-negative breast cancer and allows a complete histological response (pCR) which represents a prognostic factor for survival. . The problem for patients who are not pCR is that they are currently receiving non-personalized adjuvant systemic treatment.

The identification of biomarkers present in the residual disease would be a criterion to guide the choice of post-neoadjuvant adjuvant systemic treatment, in order to personalize it.

At the present time, there is no published study describing extensively the immune micro-environment (ME) in breast cancer, whether before or after chemotherapy, nor its modification induced by chemotherapy.

The team therefore propose to study in a retrospective and monocentric series, the modifications of the immune ME induced by a "standard" neo-adjuvant chemotherapy in patients with triple-negative CS, whether they are in complete histological response or not (n = twice 50).

The main objective of this project is to describe the changes in the immune ME of triple-negative breast cancers induced by neoadjuvant chemotherapy for all patients (in pCR or not):

* Quantification of TILs and subtypes of TILs (CD4 and CD8)
* Expression of the three immune checkpoints that are PDL1, TIM3 and LAG3
* Describe the organization of the immune system (immunostaining on the same slide of the PDL1, TIM3 and LAG3 immune checkpoints)

DETAILED DESCRIPTION:
Retrospective and monocentric translational study carried out on patients treated at the IUCT-Oncopole by neoadjuvant chemotherapy (sequential treatment FEC100 or EC100 then taxane, paclitaxel weekly for the most part) for a triple-negative CS between 2012 and 2018.

We have the microbiopsy of the primary tumor preserved in FFPE and the operating room preserved in FFPE.

We have all the clinical data for the diagnosis and monitoring of these patients, already entered into a database.

The search for a BRCA germline mutation is available in most patients if indicated for an oncogenetic consultation.

biomarkers analysis :

* TILS account according to Salgado et al. before and after neoadjuvant chemotherapy
* IHC CK5-6 and EGFR then RA if the first two are negative to characterize triple negative tumors in "basal-like" and "non-basal-like"
* IHC CD3 (labeling of T lymphocytes)
* IHC CD4, CD8 and FOXP3 before and after neoadjuvant chemotherapy
* PDL1, TIM3 and LAG3 multiplex IHC before and after neoadjuvant chemotherapy
* Labeling of tumor cells: AE1 / AE3
* Use of markings for exploratory analyzes: CD68 (macrophages), CD39 (marker of lymphocyte exhaust

ELIGIBILITY:
Inclusion Criteria:

* Samples from triple negative BC patients, patients treated by neoadjuvant chemotherapy ( FEC or EC than taxanes) Patients consent to use their samples.

Exclusion Criteria:

* Samples not available before or after neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients
Study Population: 100 samples
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Identify Change of immune ME by TILS quantification of triple-negative breast cancer induced by neoadjuvant chemotherapy for all patients | 12 months
  TILS ans substype quantification
Identify Change of immune ME by PDL1 expression of triple-negative breast cancer induced by neoadjuvant chemotherapy for all patients | 12 months
  expression of PDL1,
Identify Change of immune ME by TIM3 expression of triple-negative breast cancer induced by neoadjuvant chemotherapy for all patients | 12 months
  expression of TIM3
Identify Change of immune ME by LAG3 expression of triple-negative breast cancer induced by neoadjuvant chemotherapy for all patients | 12 months
  LAG3 expression

SECONDARY OUTCOMES:
Compare change ofTILs quantification of triple-negative breast cancer induced by neoadjuvant chemotherapy for pCR patients and those not pCR and for subtype basal-like or not basal-like | 12 months
  Quantification of TILs and subtypes TILs;
Compare change of PDL1 expression of triple-negative breast cancer induced by neoadjuvant chemotherapy for pCR patients and those not pCR and for subtype basal-like or not basal-like | 12 months
  expression of PDL1
Compare change of TIM3 expression of triple-negative breast cancer induced by neoadjuvant chemotherapy for pCR patients and those not pCR and for subtype basal-like or not basal-like | 12 months
  expression of TIM3
Compare change of LAG3 expression of triple-negative breast cancer induced by neoadjuvant chemotherapy for pCR patients and those not pCR and for subtype basal-like or not basal-like | 12 months
  expression of LAG3; organization of immune system
determination of predictive factors of TILs quantification for response to neoadjuvant chemotherapy and disease free survival | 12 months
  Correlation between TILs and TILs substypes quantification (on microbiopsy) and the histological response after neoadjuvant chemotherapy (pCR versus non pCR): determination of predictive factors for response to chemotherapy.
determination of predictive factors of PDL1 expression for response to neoadjuvant chemotherapy and disease free survival | 12 months
  Correlation between PDL1 expression on microbiopsy and the histological response after neoadjuvant chemotherapy (pCR versus non pCR): determination of predictive factors for response to chemotherapy.
determination of predictive factors of TIM3 for response to neoadjuvant chemotherapy and disease free survival | 12 months
  Correlation between TIM3 expression on microbiopsy and the histological response after neoadjuvant chemotherapy (pCR versus non pCR): determination of predictive factors for response to chemotherapy.
determination of predictive factors of LAG3 for response to neoadjuvant chemotherapy and disease free survival | 12 months
  Correlation between LAG3 expression on microbiopsy and the histological response after neoadjuvant chemotherapy (pCR versus non pCR): determination of predictive factors for response to chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut claudius regaud, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pusztai L, Foldi J, Dhawan A, DiGiovanna MP, Mamounas EP. Changing frameworks in treatment sequencing of triple-negative and HER2-positive, early-stage breast cancers. Lancet Oncol. 2019 Jul;20(7):e390-e396. doi: 10.1016/S1470-2045(19)30158-5. PMID 31267973
- [Result] Symmans WF, Peintinger F, Hatzis C, Rajan R, Kuerer H, Valero V, Assad L, Poniecka A, Hennessy B, Green M, Buzdar AU, Singletary SE, Hortobagyi GN, Pusztai L. Measurement of residual breast cancer burden to predict survival after neoadjuvant chemotherapy. J Clin Oncol. 2007 Oct 1;25(28):4414-22. doi: 10.1200/JCO.2007.10.6823. Epub 2007 Sep 4. PMID 17785706
- [Result] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Result] von Minckwitz G, Huang CS, Mano MS, Loibl S, Mamounas EP, Untch M, Wolmark N, Rastogi P, Schneeweiss A, Redondo A, Fischer HH, Jacot W, Conlin AK, Arce-Salinas C, Wapnir IL, Jackisch C, DiGiovanna MP, Fasching PA, Crown JP, Wulfing P, Shao Z, Rota Caremoli E, Wu H, Lam LH, Tesarowski D, Smitt M, Douthwaite H, Singel SM, Geyer CE Jr; KATHERINE Investigators. Trastuzumab Emtansine for Residual Invasive HER2-Positive Breast Cancer. N Engl J Med. 2019 Feb 14;380(7):617-628. doi: 10.1056/NEJMoa1814017. Epub 2018 Dec 5. PMID 30516102
- [Result] Masuda N, Lee SJ, Ohtani S, Im YH, Lee ES, Yokota I, Kuroi K, Im SA, Park BW, Kim SB, Yanagita Y, Ohno S, Takao S, Aogi K, Iwata H, Jeong J, Kim A, Park KH, Sasano H, Ohashi Y, Toi M. Adjuvant Capecitabine for Breast Cancer after Preoperative Chemotherapy. N Engl J Med. 2017 Jun 1;376(22):2147-2159. doi: 10.1056/NEJMoa1612645. PMID 28564564
- [Result] Adams S, Gray RJ, Demaria S, Goldstein L, Perez EA, Shulman LN, Martino S, Wang M, Jones VE, Saphner TJ, Wolff AC, Wood WC, Davidson NE, Sledge GW, Sparano JA, Badve SS. Prognostic value of tumor-infiltrating lymphocytes in triple-negative breast cancers from two phase III randomized adjuvant breast cancer trials: ECOG 2197 and ECOG 1199. J Clin Oncol. 2014 Sep 20;32(27):2959-66. doi: 10.1200/JCO.2013.55.0491. PMID 25071121
- [Result] Loi S, Sirtaine N, Piette F, Salgado R, Viale G, Van Eenoo F, Rouas G, Francis P, Crown JP, Hitre E, de Azambuja E, Quinaux E, Di Leo A, Michiels S, Piccart MJ, Sotiriou C. Prognostic and predictive value of tumor-infiltrating lymphocytes in a phase III randomized adjuvant breast cancer trial in node-positive breast cancer comparing the addition of docetaxel to doxorubicin with doxorubicin-based chemotherapy: BIG 02-98. J Clin Oncol. 2013 Mar 1;31(7):860-7. doi: 10.1200/JCO.2011.41.0902. Epub 2013 Jan 22. PMID 23341518
- [Result] Loi S, Drubay D, Adams S, Pruneri G, Francis PA, Lacroix-Triki M, Joensuu H, Dieci MV, Badve S, Demaria S, Gray R, Munzone E, Lemonnier J, Sotiriou C, Piccart MJ, Kellokumpu-Lehtinen PL, Vingiani A, Gray K, Andre F, Denkert C, Salgado R, Michiels S. Tumor-Infiltrating Lymphocytes and Prognosis: A Pooled Individual Patient Analysis of Early-Stage Triple-Negative Breast Cancers. J Clin Oncol. 2019 Mar 1;37(7):559-569. doi: 10.1200/JCO.18.01010. Epub 2019 Jan 16. PMID 30650045
- [Result] DeNardo DG, Barreto JB, Andreu P, Vasquez L, Tawfik D, Kolhatkar N, Coussens LM. CD4(+) T cells regulate pulmonary metastasis of mammary carcinomas by enhancing protumor properties of macrophages. Cancer Cell. 2009 Aug 4;16(2):91-102. doi: 10.1016/j.ccr.2009.06.018. PMID 19647220
- [Result] Mahmoud SM, Paish EC, Powe DG, Macmillan RD, Grainge MJ, Lee AH, Ellis IO, Green AR. Tumor-infiltrating CD8+ lymphocytes predict clinical outcome in breast cancer. J Clin Oncol. 2011 May 20;29(15):1949-55. doi: 10.1200/JCO.2010.30.5037. Epub 2011 Apr 11. PMID 21483002
- [Result] Mahmoud SM, Lee AH, Paish EC, Macmillan RD, Ellis IO, Green AR. The prognostic significance of B lymphocytes in invasive carcinoma of the breast. Breast Cancer Res Treat. 2012 Apr;132(2):545-53. doi: 10.1007/s10549-011-1620-1. Epub 2011 Jun 14. PMID 21671016
- [Result] Gu-Trantien C, Loi S, Garaud S, Equeter C, Libin M, de Wind A, Ravoet M, Le Buanec H, Sibille C, Manfouo-Foutsop G, Veys I, Haibe-Kains B, Singhal SK, Michiels S, Rothe F, Salgado R, Duvillier H, Ignatiadis M, Desmedt C, Bron D, Larsimont D, Piccart M, Sotiriou C, Willard-Gallo K. CD4(+) follicular helper T cell infiltration predicts breast cancer survival. J Clin Invest. 2013 Jul;123(7):2873-92. doi: 10.1172/JCI67428. Epub 2013 Jun 17. PMID 23778140
- [Result] Mamessier E, Sylvain A, Thibult ML, Houvenaeghel G, Jacquemier J, Castellano R, Goncalves A, Andre P, Romagne F, Thibault G, Viens P, Birnbaum D, Bertucci F, Moretta A, Olive D. Human breast cancer cells enhance self tolerance by promoting evasion from NK cell antitumor immunity. J Clin Invest. 2011 Sep;121(9):3609-22. doi: 10.1172/JCI45816. Epub 2011 Aug 15. PMID 21841316
- [Result] Bates GJ, Fox SB, Han C, Leek RD, Garcia JF, Harris AL, Banham AH. Quantification of regulatory T cells enables the identification of high-risk breast cancer patients and those at risk of late relapse. J Clin Oncol. 2006 Dec 1;24(34):5373-80. doi: 10.1200/JCO.2006.05.9584. PMID 17135638
- [Result] Mahmoud SM, Paish EC, Powe DG, Macmillan RD, Lee AH, Ellis IO, Green AR. An evaluation of the clinical significance of FOXP3+ infiltrating cells in human breast cancer. Breast Cancer Res Treat. 2011 May;127(1):99-108. doi: 10.1007/s10549-010-0987-8. Epub 2010 Jun 17. PMID 20556505
- [Result] Thibaudin M, Chaix M, Boidot R, Vegran F, Derangere V, Limagne E, Berger H, Ladoire S, Apetoh L, Ghiringhelli F. Human ectonucleotidase-expressing CD25high Th17 cells accumulate in breast cancer tumors and exert immunosuppressive functions. Oncoimmunology. 2015 Jul 6;5(1):e1055444. doi: 10.1080/2162402X.2015.1055444. eCollection 2016. PMID 26942062
- [Result] Mahmoud SM, Lee AH, Paish EC, Macmillan RD, Ellis IO, Green AR. Tumour-infiltrating macrophages and clinical outcome in breast cancer. J Clin Pathol. 2012 Feb;65(2):159-63. doi: 10.1136/jclinpath-2011-200355. Epub 2011 Nov 2. PMID 22049225
- [Result] Dieci MV, Criscitiello C, Goubar A, Viale G, Conte P, Guarneri V, Ficarra G, Mathieu MC, Delaloge S, Curigliano G, Andre F. Prognostic value of tumor-infiltrating lymphocytes on residual disease after primary chemotherapy for triple-negative breast cancer: a retrospective multicenter study. Ann Oncol. 2014 Mar;25(3):611-618. doi: 10.1093/annonc/mdt556. Epub 2014 Jan 8. PMID 24401929
- [Result] Miyashita M, Sasano H, Tamaki K, Hirakawa H, Takahashi Y, Nakagawa S, Watanabe G, Tada H, Suzuki A, Ohuchi N, Ishida T. Prognostic significance of tumor-infiltrating CD8+ and FOXP3+ lymphocytes in residual tumors and alterations in these parameters after neoadjuvant chemotherapy in triple-negative breast cancer: a retrospective multicenter study. Breast Cancer Res. 2015 Sep 4;17(1):124. doi: 10.1186/s13058-015-0632-x. PMID 26341640
- [Result] Loi S, Dushyanthen S, Beavis PA, Salgado R, Denkert C, Savas P, Combs S, Rimm DL, Giltnane JM, Estrada MV, Sanchez V, Sanders ME, Cook RS, Pilkinton MA, Mallal SA, Wang K, Miller VA, Stephens PJ, Yelensky R, Doimi FD, Gomez H, Ryzhov SV, Darcy PK, Arteaga CL, Balko JM. RAS/MAPK Activation Is Associated with Reduced Tumor-Infiltrating Lymphocytes in Triple-Negative Breast Cancer: Therapeutic Cooperation Between MEK and PD-1/PD-L1 Immune Checkpoint Inhibitors. Clin Cancer Res. 2016 Mar 15;22(6):1499-509. doi: 10.1158/1078-0432.CCR-15-1125. Epub 2015 Oct 29. PMID 26515496
- [Result] Denkert C, Loibl S, Noske A, Roller M, Muller BM, Komor M, Budczies J, Darb-Esfahani S, Kronenwett R, Hanusch C, von Torne C, Weichert W, Engels K, Solbach C, Schrader I, Dietel M, von Minckwitz G. Tumor-associated lymphocytes as an independent predictor of response to neoadjuvant chemotherapy in breast cancer. J Clin Oncol. 2010 Jan 1;28(1):105-13. doi: 10.1200/JCO.2009.23.7370. Epub 2009 Nov 16. PMID 19917869
- [Result] Denkert C, von Minckwitz G, Brase JC, Sinn BV, Gade S, Kronenwett R, Pfitzner BM, Salat C, Loi S, Schmitt WD, Schem C, Fisch K, Darb-Esfahani S, Mehta K, Sotiriou C, Wienert S, Klare P, Andre F, Klauschen F, Blohmer JU, Krappmann K, Schmidt M, Tesch H, Kummel S, Sinn P, Jackisch C, Dietel M, Reimer T, Untch M, Loibl S. Tumor-infiltrating lymphocytes and response to neoadjuvant chemotherapy with or without carboplatin in human epidermal growth factor receptor 2-positive and triple-negative primary breast cancers. J Clin Oncol. 2015 Mar 20;33(9):983-91. doi: 10.1200/JCO.2014.58.1967. Epub 2014 Dec 22. PMID 25534375
- [Result] Ladoire S, Mignot G, Dabakuyo S, Arnould L, Apetoh L, Rebe C, Coudert B, Martin F, Bizollon MH, Vanoli A, Coutant C, Fumoleau P, Bonnetain F, Ghiringhelli F. In situ immune response after neoadjuvant chemotherapy for breast cancer predicts survival. J Pathol. 2011 Jul;224(3):389-400. doi: 10.1002/path.2866. Epub 2011 Mar 25. PMID 21437909
- [Result] Burugu S, Gao D, Leung S, Chia SK, Nielsen TO. LAG-3+ tumor infiltrating lymphocytes in breast cancer: clinical correlates and association with PD-1/PD-L1+ tumors. Ann Oncol. 2017 Dec 1;28(12):2977-2984. doi: 10.1093/annonc/mdx557. PMID 29045526
- [Result] Salgado R, Denkert C, Demaria S, Sirtaine N, Klauschen F, Pruneri G, Wienert S, Van den Eynden G, Baehner FL, Penault-Llorca F, Perez EA, Thompson EA, Symmans WF, Richardson AL, Brock J, Criscitiello C, Bailey H, Ignatiadis M, Floris G, Sparano J, Kos Z, Nielsen T, Rimm DL, Allison KH, Reis-Filho JS, Loibl S, Sotiriou C, Viale G, Badve S, Adams S, Willard-Gallo K, Loi S; International TILs Working Group 2014. The evaluation of tumor-infiltrating lymphocytes (TILs) in breast cancer: recommendations by an International TILs Working Group 2014. Ann Oncol. 2015 Feb;26(2):259-71. doi: 10.1093/annonc/mdu450. Epub 2014 Sep 11. PMID 25214542